CLINICAL TRIAL: NCT04716634
Title: A Multicenter, Open-label Phase 2 Study to Evaluate the Efficacy and Safety of Tislelizumab in Combination With Fruquintinib in Patients With Selected Solid Tumors
Brief Title: Efficacy and Safety of Tislelizumab in Combination With Fruquintinib in Participants With Selected Solid Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: BeiGene (Industry)
Collaborators: Hutchison Medipharma Limited (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BGB-A317-fruquintinib-201; CTR20211070 (Other: ChinaDrugTrials)
Record Dates: First submitted 2021-01-13; First posted 2021-01-20 (Actual); Results first posted 2025-03-25 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Advanced Solid Tumors
Keywords: Solid tumors
MeSH Terms: interventions — tislelizumab; HMPL-013

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Gastric Cancer (GC): Tislelizumab and Fruquintinib (Experimental): Participants with advanced or metastatic, unresectable GC received fruquintinib 5 milligrams (mg) daily (3 weeks receiving fruquintinib followed by 1 week off) in combination with tislelizumab 300 mg intravenously on Day 1 of every 4-week cycle (each cycle of 28-days) until disease progression, unacceptable toxicity, or withdrawal for other reasons, whichever occurred first.
  Interventions: Drug: Tislelizumab; Drug: Fruquintinib
- Colorectal Cancer (CRC): Tislelizumab and Fruquintinib (Experimental): Participants with advanced or metastatic, unresectable CRC received fruquintinib 5 mg daily (3 weeks receiving fruquintinib followed by 1 week off) in combination with tislelizumab 300 mg intravenously on Day 1 of every 4-week cycle (each cycle of 28-days) until disease progression, unacceptable toxicity, or withdrawal for other reasons, whichever occurred first.
  Interventions: Drug: Tislelizumab; Drug: Fruquintinib
- PD-L1 + NSCLC: Tislelizumab and Fruquintinib (Experimental): Participants with programmed cell death protein ligand-1 (PD-L1) expression, and advanced or metastatic, unresectable non-small cell lung cancer (NSCLC) received fruquintinib 5 mg daily (3 weeks receiving fruquintinib followed by 1 week off) in combination with tislelizumab 300 mg intravenously on Day 1 of every 4-week cycle (each cycle of 28-days) until disease progression, unacceptable toxicity, or withdrawal for other reasons, whichever occurred first.
  Interventions: Drug: Tislelizumab; Drug: Fruquintinib

INTERVENTIONS:
Drug: Tislelizumab — Tislelizumab is a humanized, immunoglobulin G4 (IgG4)-variant monoclonal antibody against PD 1.
  Other Names: BGB-A317
Drug: Fruquintinib — Fruquintinib is a potent, oral VEGFR tyrosine kinase inhibitor (TKI)
  Other Names: HMPL-013

SUMMARY:
This was an open label, multicenter, Phase 2 study designed to assess the efficacy and safety of tislelizumab in combination with fruquintinib in participants with advanced or metastatic, unresectable gastric cancer (GC), or colorectal cancer (CRC) or non-small cell lung cancer (NSCLC). The study was conducted in 2 parts. Part 1 was the safety run-in stage to determine dose-limiting toxicity (DLT) and recommended Phase 2 dose (RP2D). Part 2 assessed the preliminary efficacy of tislelizumab in combination with fruquintinib in participants as measured by the overall response rate (ORR) and other efficacy and safety profiles.

DETAILED DESCRIPTION:
This was an open label, multicenter, Phase 2 study designed to assess the efficacy and safety of tislelizumab in combination with fruquintinib in patients with advanced or metastatic, unresectable GC, and CRC or NSCLC. The study was conducted in 2 parts.

Part 1 of the study was the safety run-in stage which assessed dose-limiting toxicities (DLTs) and RP2D. Part 2 began at RP2D. Participants enrolled in Part 1 at RP2D were counted towards Part 2; up to approximately 30 patients per cohort were enrolled at RP2D.

The primary outcome measure of the study was ORR as assessed by the investigator as per response evaluation criteria in solid tumors (RECIST) version (v) 1.1. Tislelizumab and fruquintinib were administered until disease progression, intolerable toxicity, death, withdrawal of consent or until the study terminates.

ELIGIBILITY:
Key Inclusion Criteria:

1. Signed informed consent form (ICF) and able to comply with study requirements.
2. At least 1 measurable lesion as defined by RECIST v1.1
3. Tumor tissue (archival tumor tissues as formalin-fixed paraffin-embedded blocks or approximately 15 unstained slides) for central laboratory assessment
4. Eastern Cooperative Oncology Group (ECOG) Performance Status less than or equal to (<=) 1
5. Histologically or cytologically confirmed, advanced or metastatic, unresectable adenocarcinoma of gastric or esophagogastric junction or colon or rectum, and histologically or cytologically confirmed, locally advanced (Stage IIIB) not amenable to curative surgery or radiotherapy, or metastatic (Stage IV) NSCLC

Key Exclusion Criteria:

1. Had at screening any central nervous system metastasis and/or leptomeningeal disease
2. Prior therapy targeting CTLA-4, PD-1, PD-L1 or programmed cell death protein ligand-2 (PD-L2) or any other antibody or drug specifically targeting T-cell costimulation or checkpoint pathways
3. Prior treatment with VEGFR-TKI or anti-VEGFR antibody (eg, ramucirumab)
4. Received more than 1 line of systemic treatment for advanced or metastatic, unresectable adenocarcinoma of gastric or esophagogastric junction, or more than 2 lines of systemic treatment for advanced or metastatic, unresectable adenocarcinoma of the colon or rectum, or prior systemic therapy for advanced or metastatic NSCLC
5. Active autoimmune diseases or history of autoimmune diseases that may relapse, or history of interstitial lung disease, noninfectious pneumonitis, or uncontrolled lung diseases including but not limited to pulmonary fibrosis, acute lung diseases, etc.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2021-04-19 (Actual); Primary Completion 2024-02-22 (Actual); Study Completion 2024-02-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jian Li, Study Director — BeiGene
Locations (13):
- China (10):
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - The First Hospital of Lanzhou University, Lanzhou, Gansu
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Shandong Cancer Hospital, Jinan, Shandong
  - Liaocheng Peoples Hospital, Liaocheng, Shandong
  - Linyi Cancer Hospital, Linyi, Shandong
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality
  - Sir Run Run Shaw Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
- South Korea (3):
  - National Cancer Center, Goyang-si, Gyeonggi-do
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Asan Medical Center, Seoul, Seoul Teugbyeolsi

IPD SHARING:
Plan to Share IPD: Yes
BeiGene shares data on completed studies responsibly and provides qualified scientific and medical researchers access to data and supporting documentation for clinical trials in dossiers for medicines and indications after submission and approval in the United States, China, and Europe. Clinical trials supporting subsequent local approvals, new indications, or combination products are eligible for sharing once corresponding regulatory approvals are achieved.
  BeiGene shares data only when permitted by applicable data privacy and security laws and regulations, when it is feasible to do so without compromising the privacy of study participants, and other considerations.
  Qualified researchers with appropriate competencies who are engaged in novel scientific research may submit a request for participant-level data with a research proposal for BeiGene review. Research teams must include a biostatistician and sign a Data Sharing Agreement prior to receiving access to clinical trial data.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See plan description
Access Criteria: See plan description
URL: http://beigene.com/science/clinical-trials/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study consisted of 2 parts: Part 1 (Safety run-in) and Part 2 (Extension). Part 1 of the study with limited participants assessed dose-limiting toxicities (DLTs) and recommended Phase 2 dose (RP2D). These participants later moved to Part 2 of the study. Participant flow, baseline demographics and adverse event data were planned to be reported and analyzed for the combined Part 1 and Part 2 of study. All participants received same dose of study drugs (tislelizumab and fruquintinib).
Period: Overall Study
Arm/Group | Gastric Cancer (GC): Tislelizumab and Fruquintinib | Colorectal Cancer (CRC): Tislelizumab and Fruquintinib | PD-L1 + NSCLC: Tislelizumab and Fruquintinib
Started | 31 | 31 | 22
Completed | 2 | 3 | 7
Not Completed | 29 | 28 | 15
Not completed — Death | 24 | 24 | 8
Not completed — Closed by Sponsor | 4 | 4 | 5
Not completed — Lost to Follow-up | 1 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Analysis was performed on safety analysis set that included all participants who received at least 1 dose of study drug(s).
Groups:
- Gastric Cancer (GC): Tislelizumab and Fruquintinib: Participants with advanced or metastatic, unresectable GC received fruquintinib 5 mg daily (3 weeks receiving fruquintinib followed by 1 week off) in combination with tislelizumab 300 mg intravenously on Day 1 of every 4-week cycle (each cycle of 28-days) until disease progression, unacceptable toxicity, or withdrawal for other reasons, whichever occurred first.
- PD-L1 + NSCLC: Tislelizumab and Fruquintinib: Participants with PD-L1 expression, and advanced or metastatic, unresectable NSCLC received fruquintinib 5 mg daily (3 weeks receiving fruquintinib followed by 1 week off) in combination with tislelizumab 300 mg intravenously on Day 1 of every 4-week cycle (each cycle of 28-days) until disease progression, unacceptable toxicity, or withdrawal for other reasons, whichever occurred first.
- Total: Total of all reporting groups
Arm/Group | Gastric Cancer (GC): Tislelizumab and Fruquintinib | Colorectal Cancer (CRC): Tislelizumab and Fruquintinib | PD-L1 + NSCLC: Tislelizumab and Fruquintinib | Total
Number analyzed (Participants) | 31 | 31 | 22 | 84
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.0 (8.71) | 58.8 (7.88) | 63.5 (11.28) | 60.1 (9.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 11 | 5 | 26
  Male | 21 | 20 | 17 | 58
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 30 | 31 | 22 | 83
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0
  More than one race | 1 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Number of Participants With Dose Limiting Toxicities (DLTs)
Description: A DLT was defined as 1 of the following toxicities (Grade 3 or 4 Hematologic or Nonhematologic toxicities) occurring during the DLT assessment window and considered by the investigator to be related to 1 or more study drugs. All toxicities or adverse events (AEs) were graded according to the National Cancer Institute-Common Terminology Criteria for Adverse Events version 5.0 (NCI-CTCAE v5.0).
Time Frame: Up to 28 Days
Population: Analysis was performed on the DLT evaluable analysis set that included all participants in Part 1 who received at least 85% of the assigned total dose of fruquintinib and at least 67% of the assigned total dose of tislelizumab during the DLT assessment period.
Measure: Count of Participants; unit: Participants
Groups:
- Tislelizumab and Fruquintinib: All participants received the full dose of fruquintinib 5 mg daily (3 weeks receiving fruquintinib followed by 1 week off) in combination with tislelizumab 300 mg intravenously on Day 1 of every 4-week cycle (each cycle of 28-days) until disease progression, unacceptable toxicity, or withdrawal for other reasons, whichever occurred first.
Arm/Group | Tislelizumab and Fruquintinib
Number analyzed (Participants) | 6
Participants | 0

2. Primary Outcome: Part 1: Recommended Phase 2 Dose (RP2D)
Description: RP2D for Part 2 was determined by evaluating safety and DLTs in Part 1 participants.
Time Frame: Up to 28 Days
Population: Analysis was performed on the DLT evaluable analysis set.
Measure: Number; unit: milligrams (mg) per day
Arm/Group | Tislelizumab and Fruquintinib
Number analyzed (Participants) | 6
milligrams (mg) per day | 5.0

3. Primary Outcome: Objective Response Rate (ORR) as Assessed by the Investigator Based on Response Evaluation Criteria in Solid Tumors (RECIST) Version (v)1.1
Description: ORR was defined as the percentage of participants achieving a best overall response (BOR) of complete response (CR) or partial response (PR). Per RECIST v1.1., CR was defined as disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to less than (<) 10 millimeters (mm). PR was defined as at least a 30 percent (%) decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: From date of randomization until the date of first documented progression or death from any cause, whichever came first (up to 2 years and 9 months)
Population: Analysis was performed on the safety analysis set which included all participants who received at least 1 dose of study drug(s).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Gastric Cancer (GC): Tislelizumab and Fruquintinib | Colorectal Cancer (CRC): Tislelizumab and Fruquintinib | PD-L1 + NSCLC: Tislelizumab and Fruquintinib
Number analyzed (Participants) | 31 | 31 | 22
percentage of participants | 12.9 [3.6 to 29.8] | 9.7 [2.0 to 25.8] | 40.9 [20.7 to 63.6]

4. Secondary Outcome: Progression-Free Survival (PFS) as Assessed by Investigator Based on RECIST v1.1
Description: PFS was defined as the time from the date of the first dose of study drug(s) to the date of the confirmed documentation of progressive disease (PD) or death, whichever occurs first. Median PFS was estimated using the Kaplan-Meier method. Per RECIST v1.1, PD was defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study.
Time Frame: From date of first dose of study drug until the date of first documented progression or death from any cause, whichever came first (up to 2 years and 9 months)
Population: Analysis was performed on the safety analysis set.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Gastric Cancer (GC): Tislelizumab and Fruquintinib | Colorectal Cancer (CRC): Tislelizumab and Fruquintinib | PD-L1 + NSCLC: Tislelizumab and Fruquintinib
Number analyzed (Participants) | 31 | 31 | 22
months | 4.6 [3.4 to 7.4] | 4.6 [3.6 to 7.2] | 15.6 [1.8 to NA] — The upper limit of 95% confidence interval (CI) could not be calculated due to fewer number of participants with events.

5. Secondary Outcome: Disease Control Rate (DCR) as Assessed by the Investigator Based on RECIST v1.1
Description: DCR was defined as the percentage of participants whose best overall response is CR, PR, or stable disease (SD) as assessed by investigator as per RECIST v1.1. Per RECIST v1.1., CR was defined as disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm. PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. SD: Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study.
Time Frame: as for outcome 3
Population: Analysis was performed on the safety analysis set.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Gastric Cancer (GC): Tislelizumab and Fruquintinib | Colorectal Cancer (CRC): Tislelizumab and Fruquintinib | PD-L1 + NSCLC: Tislelizumab and Fruquintinib
Number analyzed (Participants) | 31 | 31 | 22
percentage of participants | 74.2 [55.4 to 88.1] | 74.2 [55.4 to 88.1] | 68.2 [45.1 to 86.1]

6. Secondary Outcome: Clinical Benefit Rate (CBR) as Assessed by the Investigator Based on RECIST v1.1
Description: CBR was defined as the percentage of participants whose best overall response is CR, PR, or durable stable disease (SD) as assessed by the investigator per RECIST v1.1. Per RECIST v1.1., CR was defined as disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm. PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. SD: Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study.
Time Frame: as for outcome 3
Population: Analysis was performed on the safety analysis set.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Gastric Cancer (GC): Tislelizumab and Fruquintinib | Colorectal Cancer (CRC): Tislelizumab and Fruquintinib | PD-L1 + NSCLC: Tislelizumab and Fruquintinib
Number analyzed (Participants) | 31 | 31 | 22
percentage of participants | 32.3 [16.7 to 51.4] | 38.7 [21.8 to 57.8] | 59.1 [36.4 to 79.3]

7. Secondary Outcome: Duration of Response (DOR) as Assessed by The Investigator Based on RECIST v1.1
Description: DOR was defined as the time from the first occurrence of documented objective response to the time of progression as assessed by investigator per RECIST v1.1 or death from any cause, whichever occurs first. Median DOR was estimated using the Kaplan-Meier method.
Time Frame: From the first objective response to the date of first documentation of disease progression or death, whichever occurs first (up to 2 years and 9 months)
Population: Analysis was performed using participants in the safety analysis set with an objective response.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Gastric Cancer (GC): Tislelizumab and Fruquintinib | Colorectal Cancer (CRC): Tislelizumab and Fruquintinib | PD-L1 + NSCLC: Tislelizumab and Fruquintinib
Number analyzed (Participants) | 4 | 3 | 9
months | NA [5.6 to NA] — Median and the upper limit of 95% CI could not be calculated due to fewer number of participants with events. | 11.9 [3.7 to NA] — The upper limit of 95% CI could not be calculated due to fewer number of participants with events. | NA [7.7 to NA] — Median and the upper limit of 95% CI could not be calculated due to fewer number of participants with events.

8. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from the date of first dose to the date of death due to any cause. Median OS was estimated using the Kaplan-Meier method.
Time Frame: From the first dose of the study treatment to date of death from any cause (up to 2 years and 9 months)
Population: Analysis was performed on the safety analysis set.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Gastric Cancer (GC): Tislelizumab and Fruquintinib | Colorectal Cancer (CRC): Tislelizumab and Fruquintinib | PD-L1 + NSCLC: Tislelizumab and Fruquintinib
Number analyzed (Participants) | 31 | 31 | 22
months | 10.5 [5.2 to 14.6] | 10.0 [4.7 to 15.2] | NA [6.0 to NA] — Median and the upper limit of 95% CI could not be calculated due to fewer number of participants with events.

9. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Serious TEAEs, Grade 3 or Higher TEAEs, TEAEs Leading to Death, TEAEs Related to Tislelizumab, TEAEs Related to Fruquintinib
Description: A TEAE was defined as an AE that had an onset date or a worsening in severity from baseline (pre-treatment) on or after the first dose of study drug(s) and up to 30 days following study drug(s) discontinuation or initiation of new anticancer therapy, whichever occurred first determined according to NCI-CTCAE v5.0. Treatment emergent serious Adverse Events (TESAEs): any untoward medical occurrence at any dose: resulted in death; was life threatening; required prolong inpatient hospitalization; resulted in persistent or significant disability/incapacity; resulted in a congenital anomaly/birth defect or was considered a significant medical event by the investigator. AEs were graded for severity using NCI-CTCAE v5.0, where Grade 1: Mild; Grade 2: Moderate; Grade 3: Severe; Grade 4 - Life-threatening consequences; and Grade 5: Death related to AE. The TEAEs leading to death in this data table exclude death due to disease under study.
Time Frame: From the date of the first dose of study drug up to 30 days after the last dose of study drug; up to approximately 2 years and 5 months.
Population: Analysis was performed on the safety analysis set.
Measure: Count of Participants; unit: Participants
Arm/Group | Gastric Cancer (GC): Tislelizumab and Fruquintinib | Colorectal Cancer (CRC): Tislelizumab and Fruquintinib | PD-L1 + NSCLC: Tislelizumab and Fruquintinib
Number analyzed (Participants) | 31 | 31 | 22
Participants
  TEAEs | 30 | 31 | 22
  TESAEs | 13 | 14 | 13
  Grade 3 or Higher TEAEs | 18 | 21 | 18
  TEAEs Leading to Death | 3 | 0 | 1
  TEAEs Related to Tislelizumab | 20 | 22 | 16
  TEAEs Related to Fruquintinib | 25 | 26 | 19

ADVERSE EVENTS:
Time Frame: All-cause mortality data was collected through the end of study, that is, up to 2 years 9 months. Adverse event data was collected from the date of the first dose of study drug up to 30 days after the last dose of study drug (up to approximately 2 years and 5 months).
Arm/Group | Gastric Cancer (GC): Tislelizumab and Fruquintinib | Colorectal Cancer (CRC): Tislelizumab and Fruquintinib | PD-L1 + NSCLC: Tislelizumab and Fruquintinib
All-Cause Mortality (participants affected / at risk) | 24/31 | 24/31 | 8/22
Serious Adverse Events (participants affected / at risk) | 13/31 | 14/31 | 13/22
Other Adverse Events (participants affected / at risk) | 28/31 | 29/31 | 19/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gastric Cancer (GC): Tislelizumab and Fruquintinib (N=31) | Colorectal Cancer (CRC): Tislelizumab and Fruquintinib (N=31) | PD-L1 + NSCLC: Tislelizumab and Fruquintinib (N=22)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Immune-mediated myocarditis (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Ventricular arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Hypopituitarism (Endocrine disorders) | 0 (0) | 0 (0) | 2 (2)
Retinal artery occlusion (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Enterovesical fistula (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastric haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Impaired gastric emptying (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Intestinal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Large intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Asthenia (General disorders) | 1 (1) | 0 (0) | 0 (0)
Death (General disorders) | 3 (3) | 0 (0) | 2 (2)
General physical health deterioration (General disorders) | 2 (2) | 3 (3) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Biliary obstruction (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Gallbladder obstruction (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 2 (2) | 0 (0) | 0 (0)
Immune-mediated hepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 1 (1)
Multisystem inflammatory syndrome (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Biliary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Diabetic ketosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Gingival cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Ureterolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Prostatic obstruction (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dermatitis exfoliative (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gastric Cancer (GC): Tislelizumab and Fruquintinib (N=31) | Colorectal Cancer (CRC): Tislelizumab and Fruquintinib (N=31) | PD-L1 + NSCLC: Tislelizumab and Fruquintinib (N=22)
Anaemia (Blood and lymphatic system disorders) | 10 (11) | 6 (8) | 4 (6)
Coagulopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 3 (3) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Atrioventricular block first degree (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Hypertrophic cardiomyopathy (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 2 (2) | 0 (0) | 1 (1)
Hypophysitis (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
Hypopituitarism (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 7 (7) | 10 (10) | 4 (5)
Thyroid disorder (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 5 (6) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Angular cheilitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 0 (0) | 3 (7) | 0 (0)
Chronic gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 2 (3) | 10 (15) | 4 (12)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Duodenogastric reflux (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Eructation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gingival pain (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0)
Gingival swelling (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (3) | 3 (4) | 2 (4)
Periodontal disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 5 (5) | 3 (3)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 4 (4) | 4 (7) | 0 (0)
Asthenia (General disorders) | 3 (28) | 1 (1) | 1 (1)
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Chills (General disorders) | 0 (0) | 1 (1) | 0 (0)
Face oedema (General disorders) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 6 (6) | 2 (2)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 1 (1)
Malaise (General disorders) | 4 (4) | 1 (2) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 1 (1)
Pain (General disorders) | 1 (1) | 1 (1) | 0 (0)
Peripheral swelling (General disorders) | 1 (2) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 6 (12) | 3 (5)
Autoimmune hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Biliary obstruction (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Asymptomatic bacteriuria (Infections and infestations) | 0 (0) | 0 (0) | 1 (2)
COVID-19 (Infections and infestations) | 1 (1) | 1 (1) | 3 (3)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Chronic sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Cystitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gingivitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (2)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (2) | 0 (0) | 0 (0)
Oral infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pericoronitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 2 (2)
Pneumonia aspiration (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Rash pustular (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Suspected COVID-19 (Infections and infestations) | 0 (0) | 1 (2) | 1 (2)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0)
Skeletal injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 2 (2) | 0 (0)
Alanine aminotransferase increased (Investigations) | 2 (2) | 5 (8) | 3 (4)
Alpha hydroxybutyrate dehydrogenase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 4 (4) | 7 (10) | 3 (4)
Bilirubin conjugated increased (Investigations) | 1 (1) | 1 (1) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 2 (3) | 4 (6)
Blood bilirubin increased (Investigations) | 2 (2) | 5 (5) | 4 (7)
Blood bilirubin unconjugated increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood chloride decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood cholesterol increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood corticotrophin decreased (Investigations) | 1 (1) | 0 (0) | 1 (1)
Blood creatine phosphokinase MB increased (Investigations) | 0 (0) | 1 (1) | 3 (5)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 3 (5) | 1 (1) | 2 (6)
Blood fibrinogen decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood glucose increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood lactate dehydrogenase increased (Investigations) | 1 (1) | 0 (0) | 3 (4)
Blood thyroid stimulating hormone increased (Investigations) | 2 (3) | 2 (2) | 3 (5)
Blood uric acid increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 2 (2) | 2 (3) | 2 (4)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Myocardial necrosis marker increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 5 (14) | 2 (10) | 3 (4)
Neutrophil count increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Occult blood positive (Investigations) | 1 (1) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 5 (10) | 3 (6) | 4 (6)
Protein total decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Protein urine present (Investigations) | 0 (0) | 0 (0) | 1 (1)
SARS-CoV-2 test positive (Investigations) | 3 (8) | 1 (1) | 3 (3)
Urinary occult blood positive (Investigations) | 0 (0) | 0 (0) | 1 (1)
Urobilinogen urine increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 11 (12) | 3 (3) | 3 (3)
Weight increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
White blood cell count decreased (Investigations) | 7 (23) | 1 (2) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 5 (6) | 6 (9) | 4 (5)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 2 (2)
Electrolyte imbalance (Metabolism and nutrition disorders) | 2 (2) | 2 (2) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 2 (3)
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (2)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (3)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 10 (14) | 4 (4) | 9 (13)
Hypocalcaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Hypochloraemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 6 (15) | 0 (0) | 3 (10)
Hyponatraemia (Metabolism and nutrition disorders) | 4 (5) | 1 (1) | 4 (4)
Hypoproteinaemia (Metabolism and nutrition disorders) | 1 (3) | 1 (1) | 1 (1)
Hypovolaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3) | 2 (2)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Muscle fatigue (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (5) | 3 (4) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0)
Altered state of consciousness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (3)
Headache (Nervous system disorders) | 0 (0) | 3 (3) | 2 (2)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 1 (2) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1)
Albuminuria (Renal and urinary disorders) | 1 (2) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 1 (1) | 3 (5)
Proteinuria (Renal and urinary disorders) | 7 (7) | 13 (18) | 7 (17)
Urethritis noninfective (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Gynaecomastia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 2 (3) | 0 (0)
Prostatic obstruction (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Uterine disorder (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 6 (6)
Diaphragmatic spasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Laryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (3)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 0 (0)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 (1) | 7 (10) | 3 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (3) | 3 (4)
Rash (Skin and subcutaneous tissue disorders) | 1 (2) | 1 (1) | 2 (2)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 7 (7) | 6 (6) | 5 (5)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
BeiGene has 18 months from the end of the study at all sites to publish overall study results. After the 1st multi-site publication or the expiration of publication period, Investigators are free to publish/present the results of the study. Investigators must submit all draft publications/presentations to us for review 60 days prior to the planned publication/presentation date. BeiGene may request deletion of its confidential information & may request a further delay to protect its IP rights.

DOCUMENTS (2):
  • Study Protocol (2020-12-16): https://cdn.clinicaltrials.gov/large-docs/34/NCT04716634/Prot_000.pdf
  • Statistical Analysis Plan (2024-02-27): https://cdn.clinicaltrials.gov/large-docs/34/NCT04716634/SAP_001.pdf